CLINICAL TRIAL: NCT06528574
Title: Incidence of Postoperative Pain After Activation of Irrigant With Apical Negative Pressure and Ultrasonics in Mandibular Molar Teeth With Irreversible Pulpitis: A Randomized Controlled Trial
Brief Title: Postoperative Pain After Activation of Irrigant
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cleveland Dental Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CDIENDO0001
Record Dates: First submitted 2024-07-18; First posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Ultrasonography

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Conventional root canal treatment (Active Comparator): Irrigation will be performed with side vented needles only
  Interventions: Device: Conventional root canal treatment
- Irrigant activation with Ultrasonic (Experimental): Final irrigant activation will be done by ultrasonic
  Interventions: Device: Ultrasonic
- Irrigant activation with negative pressure (Experimental): Final irrigant activation will be performed with apical negative pressure
  Interventions: Device: Apical negative pressure
- Irrigant activation with both Ultrasonic and negative pressure (Experimental): Final irrigation with a combination of ultrasonic and apical negative pressure using the IVAC device.
  Interventions: Device: Combined Ultrasonic and negative pressure

INTERVENTIONS:
Device: Conventional root canal treatment — Root canals will be irrigated by only side perforated needle
  Arms: Conventional root canal treatment
Device: Ultrasonic — Root canals will finally receive activation of the irrigant by the ultrasonic part of the IVAC system
  Arms: Irrigant activation with Ultrasonic
Device: Apical negative pressure — Root canals will finally receive activation of the irrigant by the negative pressure part of the IVAC system
  Arms: Irrigant activation with negative pressure
Device: Combined Ultrasonic and negative pressure — Root canals will finally receive activation of the irrigant by the IVAC system which is a combination of ultrasonic and apical negative pressure procedures.
  Arms: Irrigant activation with both Ultrasonic and negative pressure

SUMMARY:
The purpose of this research is to analyze the levels of pain after cleaning and shaping in individuals who are receiving root canal therapy using the IVAC irrigation approach, and those who are treated with ultrasonic irrigation techniques, negative pressure irrigation technique and traditional irrigation techniques.

PICOTS Question:

Does the new Dent's iVac irrigation protocol has an effect on reduction of postoperative pain

By enlisting at least 84 suitable individuals who are undergoing the identical endodontic procedure.

pain will be measures by assessing pain levels through a standardized numerical rate scale (NRS) at certain time intervals after root canal treatment, 6 hours, 12 hours, 24 hours, 48 hours, and 72 hours.

ELIGIBILITY:
Inclusion Criteria:

Males and females Age :20-50 Mandibular mature first molars with symptomatic acute pulpitis Medically free patients

Exclusion Criteria:

Pulp necrosis or apical periodontitis Periodontal disease Vertical root fracture Radiographic apical radiolucency

-

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Numerical Pain Scale (NRS) | Preoperative, 6 hours, 12 hours, 24 hours, 48 hours and 72 hour post-procedure.
  Pain will be assessed during the numerical rate scale (NRS) which has a scale from 0 to 10, where 0 is no pain while 10 is most unbearable one.

SECONDARY OUTCOMES:
Analgesics intake | 6 hours, 12 hours, 24 hours,48 hours and 72 hour post-procedure.
  The patient will be advised to take analgesics in case of unbearable pain and record this. Number of tablets and the time will be recorded
  ● The satisfaction of patients regarding the pain management intervention at the follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed A Hashem, PhD, Study Chair — Cleveland Dental Institute
Locations (1):
- Cleveland Dental Institute, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No